CLINICAL TRIAL: NCT00911118
Title: A Phase I Dose Escalation Study Using Ultra-Hypofractionated, Image-Guided, Intensity-Modulated Radiotherapy in Prostate Cancer
Brief Title: Dose Escalation Study Using Ultra-Hypofractionated, Image-Guided, Intensity-Modulated Radiotherapy in Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-035
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer; Adenocarcinoma
Keywords: prostate; radiation; 09-035
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

ARMS (1):
- Radiation (Experimental): Patients enrolled in the study will undergo image-guided, intensity-modulated radiotherapy using the same equipment, techniques, and treatment-planning procedures as currently practiced as MSKCC. MSKCC patients will have the option of continued follow-up through MSKCC's established Prostate Survivorship Clinic for an indefinite period of time, meaning patients enrolled in the protocol will be encouraged to remain at MSKCC for life-long follow-up after their treatment. The standard assessments obtained in the Survivorship Clinic will not be altered. All protocol relevant data collected at these visits through month 60 will be used for protocol analysis.
  Interventions: Radiation: Hypofractionated, image-guided, intensity-modulated external beam radiation

INTERVENTIONS:
Radiation: Hypofractionated, image-guided, intensity-modulated external beam radiation — A standard dose escalation design is utilized, with the initial treatment assigned as 6.5 Gy/fraction for five fractions to a total dose of 32.5 Gy. For any given dose tier, an initial cohort of 30 patients will be treated. However to adjust for potentially inevaluable patients who dropout prior to a full toxicity collection to assess potential DLTs enrollment of up to five additional patients per cohort can occur, per PI's discretion. Dose escalation will proceed if < 10% of the 30 patients treated per tier exhibit any dose limiting toxicity (DLT) once the entire tier cohort has a minimum follow-up of 3 months and half the tier cohort has a minimum follow-up of 6 months. Dose escalation to the next tier will occur by increasing the dose per fraction by 0.5 Gy while keeping the fraction number constant at 5, leading to a total dose increase of 2.5 Gy per dose tier.

SUMMARY:
The purpose of this study is to test the safety of a new type of IG-IMRT called "ultra-hypofractionated IG-IMRT" where a higher dose of radiation is given to the tumor during each treatment day. Since higher doses of radiation are used each day, the total number of treatment days needed to complete this type of radiation is only five instead of the 45-48 treatments currently used. Treatment takes place every other day and is complete after 2 weeks. If the patient decides to get this treatment, they will come in for 5 treatments. This is different from the 48 treatments they would get normally.

ELIGIBILITY:
Inclusion Criteria:

Eligibility is not restricted to MSKCC to confirm biopsy/diagnosis. Participating institution testing is sufficient.

* Low and intermediate risk prostate cancer patients will be eligible for this study. Risk groups will be assigned as per NCCN guidelines.
* Low risk patients will be defined as:

  * PSA < or = to 10 ng/ml and
  * Gleason score = 6 and
  * Clinical Stage < or = to T2a
* Intermediate risk patients will be defined as:

  * PSA 10-20 ng/ml or
  * Gleason score = 7 or
  * Clinical stage T2b/T2c

Additionally, patients will be required to meet the following criteria:

* Age > or = to 18
* KPS > or = to 70
* Pre-treatment endorectal coil MRI or CT (MRI preferred) at MSKCC showing no definite evidence of radiographic T3, T4, or N1 disease
* Prostate size < or = to 60 cc
* International Prostate Symptom Score < or = to 15

Exclusion Criteria:

* Prior androgen deprivation therapy for prostate cancer

  * Elective pelvic lymph node irradiation
  * KPS < 70
  * Pelvic MRI or CT (MRI preferred) evidence of radiographic T3, T4 or N1 disease
  * Presence of distant metastasis as determined by:

    o alkaline phosphatase > or = to ULN or
  * whole body bone scan positive for osseous metastases
  * Prior history of transurethral resection of the prostate
  * Prior history of chronic prostatitis
  * Prior history of urethral stricture
  * Prior history of pelvic irradiation
  * History of inflammatory bowel disease
  * Unable to give informed consent
  * Unable to complete quality of life questionnaires Abnormal complete blood count. Any of the following

    * Platelet count less than 75,000/ml
    * Hb level less than 10 gm/dl
    * WBC less than 3.5/ml
  * Abnormal renal function tests (creatinine > 1.5)

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assess the toxicity of hypofractionated radiation therapy as definitive treatment for low and intermediate risk prostate cancer. | With at least one status check visit during the course of treatment.

SECONDARY OUTCOMES:
Evaluate post-treatment PSA kinetics and incidence of PSA relapse free survival. | 1, 3, & 6 months (+/- 4 weeks) Months 6 - 36 every 6 months (+/- 4 weeks)
Evaluate pathologic response rates at 24-36 months via repeat biopsy. | 24-36 months post treatment
Evaluate the effect of treatment on sexual function. | 1, 3, & 6 months (+/- 4 weeks) Months 6 - 36 every 6 months (+/- 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Sean McBride, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York
  - Montefiore Medical Center, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Moore A, Kollmeier MA, McBride SM, Toumbacaris N, Zhang Z, Lacy-Elsayegh A, Dreyfuss A, Grossman CE, Gorovets D, Zelefsky MJ. Long-term Outcomes from a Phase 1 Dose Escalation Study Using Stereotactic Body Radiotherapy for Patients with Low- or Intermediate-risk Prostate Cancer. Eur Urol Oncol. 2024 Aug;7(4):812-820. doi: 10.1016/j.euo.2023.10.019. Epub 2023 Nov 10. PMID 37949730
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org